CLINICAL TRIAL: NCT03548493
Title: Magnesium Sulphate Versus Fentanyl as Adjuvants to Propofol Xylocaine Combination for Conscious Sedation During Chronic Subdural Haematoma Surgery. Comparative Study
Brief Title: Magnesium Sulphate Versus Fentanyl for Conscious Sedation in CSDH
Acronym: CSDH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rania Samir Fahmy, Lecturer of Anesthesia, surgical intensive care and pain mangement, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-28-2018
Record Dates: First submitted 2018-05-12; First posted 2018-06-07 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Conscious Sedation
Keywords: Magnesium sulphate; Fentanyl; Conscious sedation; chronic subdural haematoma; Propofol; Burr hole
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Magnesium Sulfate; Fentanyl; Propofol

STUDY DESIGN:
Intervention Model Description: 34 patients are randomly divided by computer designed lists and then concealed in closed envelopes into 2 equal groups:
  1. Group A (n=17) will receive magnesium sulphate adjuvant to propofol for sedation.
  2. Group B (n=17) will receive fentanyl adjuvant to propofol for sedation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium (M) group (Experimental): Magnesium (M) group (n=17) , in which magnesium sulphate is given as adjuvant to propofol for sedation
  Interventions: Drug: Magnesium sulphate; Drug: Propofol
- Fentanyl (F) group (Active Comparator): Fentanyl (F) group (n=17), in which fentanyl is given as adjuvant to propofol for sedation
  Interventions: Drug: Fentanyl; Drug: Propofol

INTERVENTIONS:
Drug: Magnesium sulphate — Magnesium sulphate will be given to the experimental group in a dose of 50mg/kg IV over 15 minutes followed by continuous infusion at 15 mg/kg/h
  Arms: Magnesium (M) group
Drug: Fentanyl — Fentanyl will be given to the active comparator group in a dose of 1 μg /kg IV bolus over 15 minutes followed by continuous infusion starting at 0.5 μg /kg/h
  Arms: Fentanyl (F) group
Drug: Propofol — In both groups Fentanyl and magnesium sulphate will be accompanied by IV propofol at a dose of 50- 150 μg /kg) bolus over 15 minutes to achieve target sedation level, that is Ramsay sedation scale (RSS) 3,if RSS afterwards does not reach 3, a supplementary bolus dose of 0.2 mg/kg propofol will be given to the patients, followed by ( 20-40 μg /kg/ min) to maintain Intraoperative level of sedation by bispectral index (BIS ) reading by 60-80%

SUMMARY:
The investigators hypothesize that magnesium sulphate owing to its analgesic and sedative properties is not inferior to fentanyl in providing conscious sedation as adjuvants to propofol and local injection of lidocaine in patients undergoing surgery for evacuation of subdural haematoma. Consequently, the investigators are testing this hypothesis by comparing the sedative and analgesic effects of magnesium sulphate versus fentanyl as adjuvants to propofol lidocaine admixture for conscious sedation in patients undergoing burr hole surgery for evacuation of subdural haematoma.

DETAILED DESCRIPTION:
Following institutional ethical committee approval, 34 patients undergoing burr-hole surgery for chronic subdural hemorrhage were included in this prospective, randomized, double-blind study.

Written informed consent were obtained from all subjects before enrollment in the study.

During the preanesthetic checkup,the operative procedure and anesthetic techniques were explained to all patients.

Upon arrival to operating theater, standard monitoring were applied to all patients and bispectral index was applied before starting the drug infusions and was used for maintenance of sedation during operation.

Subjects were randomized into 2 groups. Magnesium (M) group received Magnesium sulphate 50mg/kg IV over 15 minutes Followed by continuous infusion at 15 mg/kg/h Fentanyl (F) group received fentanyl 1 μg /kg IV bolus over 15 minutes Followed by continuous infusion starting at 0.5 μg /kg/h Loading and infusion doses of magnesium sulphate and loading doses of fentanyl were chosen from previous studies.

In both groups fentanyl and magnesium sulphate were accompanied by IV propofol at a dose of 50- 150 μg /kg/min bolus over 10 minutes to achieve target sedation level, that is, Ramsay sedation scale (RSS) 3, if RSS afterwards does not reach 3, a supplementary bolus dose of 0.2 mg/kg propofol were given to the patients, followed by ( 20-40 μg /kg/ min) to maintain Intraoperative level of sedation by bispectral index (BIS ) reading by 60-80 After achieving predefined target sedation level (RSS of 3), surgeons infiltrated the sites of the burrholes with 20 mL of a local anesthetic solution containing 10 mL of 0.5% bupivacaine and 10 mL of 2% lidocaine with adrenaline infiltrated locally at least 5 minutes before surgical incision. After burr-hole craniotomy followed by the hematoma evacuation is accomplished, the Infusion of sedatives were discontinued just after placement of the final skin suture.

Intraoperative patient's movement is defined as those likely to interfere with surgical procedure such as bending of hand and/or leg and movement of head were recorded. The first intervention is to attempt patient reassurance for 30 seconds. If movement continues then the bolus dose of propofol of 0.5 mg/kg was given and infusion dose was increased in the previously described manner till the maximum dose to regain BIS sedation score between 60-80.

If the patient starts to move again the same sequence was repeated. Induction of general anesthesia was deemed the final intervention in case satisfactory condition was not achieved within the rescue propofol.

All patients were transferred to the post-anesthesia care unit (PACU) after surgery.

The data collected are:

1. Total amount of Propofol consumption.
2. Total number of patient movements
3. The intraoperative and postoperative hemodynamic data
4. VAS (Visual analogue scale for pain) score
5. Time to first rescue analgesic
6. Adverse events
7. Surgeon satisfaction score was recorded.

Statistical analysis:

Data was analyzed using SPSS © Statistics version 23 (IBM© Corp., Armonk, NY, USA). Chi-square test (Fisher's exact test) was used to examine the relation between qualitative variables. For quantitative data, comparison between the two groups was done using independent sample t-test or Mann-Whitney test as appropriate. All tests were two-tailed. A p-value < 0.05 was considered significant.

Sample Size calculation:

A previous study reported that pre-procedure magnesium sulphate reduced the total propofol requirements to 130±19.09 mg compared to 172.8±29.09 mg with pre-procedure fentanyl. Based on these results, a sample size of 15 cases in each group was satisfactory to elicit the difference at an alpha level of 0.05 and a power of the test of 95%. The sample size was increased to 17 per group to compensate for possible dropouts.

ELIGIBILITY:
Inclusion Criteria:

* age > 50 years
* ASA (American Society of Anesthesiologists physical status) grade I to II
* Glasgow coma scale 14-15
* Unilateral chronic subdural hematoma

Exclusion Criteria:

* Hypertension (diastolic blood pressure > 160 mmHg)
* Bradycardia (<50 bpm)
* Ischemic heart disease (<6 months)
* Second- or third-degree heart block
* Long-term abuse of or addiction to alcohol, tobacco, opioids, and sedative-hypnotic drugs (>6 months)
* Allergy to study drugs
* Neuropsychiatric diseases
* Predicted difficult airway according to Ganzouri score >4.
* Patients with deviation in the surgical technique or with inadequacy of local anesthesia were excluded from the study.

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
Total amount of Propofol consumption in each group | From the start of propofol infusion after arrival to the operating room and throughout the duration of the surgery
  To measure total amount of propofol consumption from induction of conscious sedation till the end of the operation and to compare it between both groups

SECONDARY OUTCOMES:
To measure the total number of intraoperative patient's movements | From the start of the surgery and throughout the duration of the surgery
  Intraoperative patient's movement is defined as those likely to interfere with surgical procedure such as bending of hand and/or leg and movement of head
Heart rate | Arrival at the operating room, after bolus administration of drug, at skin incision, at 1,2,5,10,15 min and 10 min after skin incision, every 15 minutes intraoperative, on arrival, 5,10,15,30 min and 1 hour at the PACU
  Heart rate in beats/min
Non invasive blood pressure | Arrival at the operating room, after bolus administration of drug, at skin incision, at 1,2,5,10,15 min and 10 min after skin incision, every 15 minutes intraoperative, on arrival, 5,10,15,30 min and 1 hour at the PACU
  Systolic and diastolic blood pressure in mmhg
To assess surgeon satisfaction score | 30 minutes after the end of the surgery
  Surgeon satisfaction was assessed as follows: 1, extremely dissatisfied; 2, not satisfied but able to manage; 3, satisfied; 4, extremely satisfied.
VAS score for pain | at skin closure and at 1hr, 2 hrs. 3hrs and 6 hrs. after PACU admission.
  The pain VAS is a unidimensional measure of pain intensity, the score is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale])
Time to first rescue analgesic | During the first 24 hours in the postoperative period
  The time when the patient first requires analgesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Aini Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guzel A, Kaya S, Ozkan U, Ufuk Aluclu M, Ceviz A, Belen D. Surgical treatment of chronic subdural haematoma under monitored anaesthesia care. Swiss Med Wkly. 2008 Jul 12;138(27-28):398-403. doi: 10.4414/smw.2008.12121. PMID 18642135
- [Background] Bishnoi V, Kumar B, Bhagat H, Salunke P, Bishnoi S. Comparison of Dexmedetomidine Versus Midazolam-Fentanyl Combination for Monitored Anesthesia Care During Burr-Hole Surgery for Chronic Subdural Hematoma. J Neurosurg Anesthesiol. 2016 Apr;28(2):141-6. doi: 10.1097/ANA.0000000000000194. PMID 26018670
- [Background] Sato M, Shirakami G, Fukuda K. Comparison of general anesthesia and monitored anesthesia care in patients undergoing breast cancer surgery using a combination of ultrasound-guided thoracic paravertebral block and local infiltration anesthesia: a retrospective study. J Anesth. 2016 Apr;30(2):244-51. doi: 10.1007/s00540-015-2111-z. Epub 2015 Dec 10. PMID 26661141
- [Background] Drown MB. Integrative review utilizing dexmedetomidine as an anesthetic for monitored anesthesia care and regional anesthesia. Nurs Forum. 2011 Jul-Sep;46(3):186-94. doi: 10.1111/j.1744-6198.2011.00229.x. PMID 21806629
- [Background] David H, Shipp J. A randomized controlled trial of ketamine/propofol versus propofol alone for emergency department procedural sedation. Ann Emerg Med. 2011 May;57(5):435-41. doi: 10.1016/j.annemergmed.2010.11.025. Epub 2011 Jan 21. PMID 21256626
- [Background] Wang W, Feng L, Bai F, Zhang Z, Zhao Y, Ren C. The Safety and Efficacy of Dexmedetomidine vs. Sufentanil in Monitored Anesthesia Care during Burr-Hole Surgery for Chronic Subdural Hematoma: A Retrospective Clinical Trial. Front Pharmacol. 2016 Nov 3;7:410. doi: 10.3389/fphar.2016.00410. eCollection 2016. PMID 27857689
- [Background] Lauretti GR. Mechanisms of analgesia of intravenous lidocaine. Rev Bras Anestesiol. 2008 May-Jun;58(3):280-6. doi: 10.1590/s0034-70942008000300011. English, Portuguese. PMID 19378524
- [Background] Cizmeci P, Ozkose Z. Magnesium sulphate as an adjuvant to total intravenous anesthesia in septorhinoplasty: a randomized controlled study. Aesthetic Plast Surg. 2007 Mar-Apr;31(2):167-73. doi: 10.1007/s00266-006-0194-5. PMID 17437152
- [Background] Prontera A, Baroni S, Marudi A, Valzania F, Feletti A, Benuzzi F, Bertellini E, Pavesi G. Awake craniotomy anesthetic management using dexmedetomidine, propofol, and remifentanil. Drug Des Devel Ther. 2017 Mar 3;11:593-598. doi: 10.2147/DDDT.S124736. eCollection 2017. PMID 28424537